CLINICAL TRIAL: NCT00800631
Title: The Biomarker and Associated Cardiac Function in the Patients With Sepsis
Brief Title: The Biomarker and Cardiac Function in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chiung-Yuan Hsu/ Attending VS of Emergency Department, National Taiwan University Hospital
Other Study IDs: 200708002R
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The development and severity of sepsis induced myocardial dysfunction can be monitored from the serum biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis patients with 2 of the followings when arrival ER and treated > 6 hours:

  * BT >38℃ or<36℃
  * HR >90/min
  * RR >20/min or PaCO2 < 32 mmHg
  * WBC count >12×109/L or <4×109/L or immature form >10％

Exclusion Criteria:

* Age < 18
* Major trauma patients
* Pregnancy
* Willing to do not aggressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sepsis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- ER of National Taiwan Univeristy Hospital, Taipei, Taiwan